CLINICAL TRIAL: NCT01352130
Title: Comparative Electrocardiographic Effects of Intravenous Ondansetron and Granisetron in Patients Undergoing Surgery for Carcinoma Breast: A Prospective Single Blind Randomised Trial
Brief Title: Granisetron Versus Ondansetron: Comparative Effects on ECG, QTc
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Dr Atul P Kulkarni, Tata Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Akulkarni1
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2011-05-11 (Estimated); Status verified 2011-05

CONDITIONS: Prolonged QTc Interval
Keywords: Postoperative nausea and vomiting; Ondansetron; Granisetron; QTc interval
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Ondansetron; Granisetron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ondansetron (Active Comparator): Patients given Ondansetron
  Interventions: Drug: Ondansetron
- Granisetron (Active Comparator): Patients given Granisetron
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Ondansetron — Intravenous Ondansetron 8 mgs
  Other Names: 5HT3 antagonists
  Arms: Ondansetron
Drug: Granisetron — Intravenous Granisetron 1 mgs
  Other Names: 5HT3 antagonists
  Arms: Granisetron

SUMMARY:
Postoperative nausea and vomiting [PONV] are common and distressing symptoms after surgery performed under general anaesthesia. 5HT3 antagonists are routinely used for prevention as well as treatment of PONV. After IRB approval we compared the effects of ondansetron and granisetron on the various intervals on ECG in 70 patients undergoing elective surgery for carcinoma breast after written informed consent. The demographic data was collected. The administration of the anaesthetic was left to the discretion of the operating room staff specialist. In the Postoperative Recovery Room patients were randomised to receive 8 mgs of ondansetron or 1 mg of granisetron intravenously. Serial ECGs were recorded at 0 mins (before injection of study drug), 2 mins, 5 mins, 15mins, 1 hour and 2 hours. Pulse rate, Non-invasive blood pressure and SpO2 were also recorded. T

DETAILED DESCRIPTION:
This prospective, randomized, single blind study was conducted after our Institutional Review Board approved the study protocol, consent form and the randomization form. 70 consecutive ASA I-III patients (age18 to 60 years) undergoing breast surgery for carcinoma breast were included in the study after obtaining written informed consent. Patients refusing consent, with prolonged QTc interval, with arrhythmias or conduction defects and those with abnormal serum levels of potassium, calcium, magnesium were excluded. There was no standardized anaesthesia technique. The technique of induction of anaesthesia, maintenance and reversal of anaesthesia was left to the discretion of the staff anaesthetist in the operating theatre. The data on comorbidities, preoperative medications for the comorbidities, premedication, induction agents, analgesics, muscle relaxants and inhalation agents was collected.

Sample size calculation: A sample size calculation was performed [according to mean changes (difference of means) in QTc interval] to find out the number of patients needed to find a significant difference between the two drugs. To detect a QTc change from baseline of greater than 5 ms with α and β error of 0.05 and 0.20, respectively, and assuming an SD of QTc change of 10 ms using a one-sided test, a minimum of 35 subjects were needed in each antiemetic group.

Randomization: The patients (n= 70) were divided randomly in two groups by computer generated random numbers by the statisticians in the Clinical Research Secretariat (CRS) in our institute. Block randomization was done with blocks of 10, to allow stratification of the patients depending on whether they had received anthracycline based neoadjuvant chemotherapy. The list of randomization numbers and clinical details were maintained in the CRS.

Intervention: Once the patients arrived postoperatively in the recovery room, one of the investigators called the Clinical Research Secretariat (CRS) on phone, after completing the randomization form and gave the patient details. The Statistician allocated the drug the patient should receive which was prepared by the investigator which was either ondansetron 8 mg (Group O) or granisetron 1mg (Group G). A baseline 12 lead electrocardiogram was obtained before the drug was administered. After baseline ECG, patients in Group O were given intravenous 8 mg ondansetron and patients in group G were given 1 mg granisetron over 30 seconds. Subsequently serial 12 lead ECGs were done at 2 mins, 5 mins, 15mins, 1 hour and 2 hours. Pulse, blood pressure and SpO2 were also monitored at those intervals. Unfiltered Electrocardiograms were recorded at paper speed of 25mm/sec and at normal amplitude with a HP Vigilent Pagewriter 100TM device which automatically calculates and prints the heart rate and the duration of various ECG intervals. The investigators independently read and analyzed the ECG to confirm that the intervals obtained with the ECG machine were indeed accurate. QT and R-R intervals were measured for calculation of corrected QT (QTc) interval. The corrected QT (QTc) interval was calculated by using the formula described by Bezzet. [QTc = QT interval/√ (RR interval)]

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing breast surgery for carcinoma breast.
* Patients between ages 18 to 60 years.
* ASA I \ II \ III
* Patients weight between 40 and 70 kilograms.

Exclusion Criteria:

* Patient refusing consent
* Prophylactic anti emetic drug administration during intraoperative period
* Known case of prolonged QTc interval
* Known case decompensated cardiomyopathy
* Known case of cardiac arrhythmia or bundle branch block
* Case of congestive heart failure with left ventricular ejection fraction <40%
* Abnormal serum level of potassium, calcium, magnesium

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Effect of Granisetron and Ondansetron on QTc interval Prolongation at various time intervals after administration | 0 mins (before injection of study drug), 2 mins, 5 mins, 15mins, 1 hour and 2 hours
  Both drugs are known to prolong QTc and other ECG intervals

CONTACTS AND LOCATIONS:
Overall Officials: Atul P Kulkarni, MD Anaes, Principal Investigator — Professor
Locations (1):
- Tata Memorial Hopsital, Mumbai, Maharashtra, India

REFERENCES:
- [Derived] Ganjare A, Kulkarni AP. Comparative electrocardiographic effects of intravenous ondansetron and granisetron in patients undergoing surgery for carcinoma breast: A prospective single-blind randomised trial. Indian J Anaesth. 2013 Jan;57(1):41-5. doi: 10.4103/0019-5049.108560. PMID 23716765